CLINICAL TRIAL: NCT00935636
Title: An Evaluation of Efficacy of the GlideScope Cobalt Video Baton for Intubation on Children Weighing Less Than 10 Kilograms
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Peter Szmuk, Professor, University of Texas Southwestern Medical Center
Other Study IDs: 042009-046
Record Dates: First submitted 2009-07-02; First posted 2009-07-09 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Intubation
Keywords: Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect relevant airway data using the GlideScope Cobalt Video Baton 1 and 2 for intubation in a large cohort of neonates and infants weighing 10 kg or less.

DETAILED DESCRIPTION:
Neonates and infants requiring endotracheal intubation and in which the attending anesthesiologist decided to use the CGS-CVB will be included in this observational study. Data will be collected by one of the investigators or the research assistant/coordinator and recorded on a data sheet The data from these forms will be then entered by the investigator or research assistant/coordinator into a database maintained only for this study.

The decision of using the GS-CVB is at the discretion of the attending anesthesiologist. Consequently if consent would be required the anesthesiologist might feel compelled or biased to use the device against his will. This will also require that all possible patients's should be consented which will put a serious strain on the study personal.

ELIGIBILITY:
Inclusion Criteria:

* Neonates, infants and children scheduled for surgical procedures under general anesthesia and requiring endotracheal intubation
* Patients age 0 - 2 years
* Weight up to 10 kg
* American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* Patients at risk of pulmonary aspiration,
* Increased intracranial pressure
* Those with congenital cardiac diseases or
* Those with hemodynamic instability

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates and infants requiring endotracheal intubation under 10 kilograms and in which the attending anesthesiologist decided to use the CGS-CVB will be included in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Time to intubation | From the time the ETT enters the mouth until end-tidal carbon dioxide is detected on the monitor screen

SECONDARY OUTCOMES:
The time to laryngoscopic views, number of attempts, and the success rate | from the time the device enters the mouth until the best view is acknowledged.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szmuk, MD, Principal Investigator — UT Southwestern
Locations (1):
- Chlidren's Medical Center Dallas, Dallas, Texas, United States